CLINICAL TRIAL: NCT04569214
Title: A Comparative, Dose-Escalating, Placebo-Controlled Study of the Efficacy and Safety of PAZ320, Ingested Together With a Standard Meal on Post-Prandial Glucose and Insulin Blood Levels in Type II Diabetic Patients Treated With Metformin
Brief Title: The Efficacy and Safety of PAZ320 on PPG and Insulin Blood Levels in Type II Diabetic Patients
Acronym: PAZ320
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAZ320-003
Record Dates: First submitted 2013-11-13; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Type II Diabetes
Keywords: PAZ320; Type II diabetes; Metformin; Galactomannan
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PAZ320; galactomannan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A - Placebo Control (Placebo Comparator): 4 tablets of placebo
  Interventions: Other: Placebo
- B - PAZ320 Low Dose (Experimental): 2 tablets of PAZ320 and 2 tablet of placebo
  Interventions: Drug: PAZ320; Other: Placebo
- C - PAZ320 High Dose (Experimental): 4 tablet of PAZ320
  Interventions: Drug: PAZ320

INTERVENTIONS:
Drug: PAZ320 — Treatment arm B - 2 tablets of PAZ320 and 2 tablets of placebo, total of 4 tablets Treatment arm C - 4 tablets of PAZ320
  Other Names: Galactomannan
  Arms: B - PAZ320 Low Dose; C - PAZ320 High Dose
Other: Placebo — Treatment arm A - 4 tablets of placebo Treatment arm B - 2 tablets of PAZ320 and 2 tablets of placebo, total of 4 tablets
  Arms: A - Placebo Control; B - PAZ320 Low Dose

SUMMARY:
The purpose of this study is to test the efficacy of PAZ320 in diabetic patients.

DETAILED DESCRIPTION:
The purpose of the present clinical study is to test the efficacy of two doses of PAZ320 in diabetic patients already on treatment with metformin, in order to assess and quantify its effect on postprandial glucose and insulin levels after a standard meal composed of rice, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type II diabetes since at least one year, not presenting any complications of their disease.
2. Patients under treatment with Metformin up to 3g/day, given twice or three times daily. Metformin doses should not exceed 3g/day, and should be well tolerated by the patients, its dose should have been stable for the last 3 months before inclusion in the study. Metformin should be taken in the morning of the visit only after the test meal is taken. The next doses of metformin will be taken with meals after the visit, in the habitual order the patient is used to take. The patients should not stop taking metformin during the study, but continue as usual, except that in the mornings of the visits, as the patients arrive in fasting conditions, metformin should be taken after the test meal. If a concomitant combination with an oral anti diabetic agent is given, because of elevated HbA1c levels, it should be taken together with metformin after the test meal.
3. Age - between 35 and 65, male and female.
4. Females should not be pregnant or breast feeding, women of child bearing potential should guarantee anti-contraceptive measures.
5. BMI (body mass index) - between 25 and 32.
6. Patients with glycated hemoglobin (HbA1c) lower than 9%, and higher than 6.5%, HbA1c will be determined in the first visit.
7. Patients who are able to collaborate during the entire duration of the study.

Exclusion Criteria:

1. Patients with other underlying diseases, such as cardiovascular disease, renal disease, peripheral vascular disease or any condition considered to be a complication of diabetes, should be excluded from this study.
2. Patients treated with insulin subcutaneous injections or with GLP-1 agonists, or by alpha-glucosidase inhibitors or by glinides should not be included in the study.
3. HbA1c higher than 9%, or lower than 6.5%
4. Women who are either pregnant or lactating
5. Participation in another clinical study in the month preceding recruitment into the study.
6. Patients who cannot guarantee compliance.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Assess the PAZ320 effect on postprandial blood glucose levels in type II diabetic patients. | 2 weeks
  The extent and duration of PAZ320 effect on postprandial blood glucose levels in type II diabetic patients will be assessed under treatment with metformin, over 4 hours after the intake of a standard meal, using an implanted continuous glucose monitoring device.

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 2 weeks
  The secondary safety endpoint is number subjects with occurrences of following AEs: injury, surgery, accidents, or illnesses, and significant abnormalities in clinical laboratory values, psychological testing, or physical examination findings. In cases of surgical or diagnostic procedures, the condition/illness leading to such a procedure will be considered as the AE rather than the procedure itself.

CONTACTS AND LOCATIONS:
Overall Officials: LOÏK GEFFRAY, MD, Principal Investigator — Department Of Internal Medicine, Infectious Diseases And Diabetology Hopital Robert Bisson (Lisieux) Lisieux, Normandy, France
Locations (1):
- Department of Internal Medicine, Infectious Diseases and Diabetology Hopital Robert Bisson (Lisieux), Lisieux, Normandy, France